CLINICAL TRIAL: NCT01989468
Title: A Phase III, Randomized, Double-blind, Placebo-controlled Multicenter Study of Subcutaneous Secukinumab in Autoinjectors, to Demonstrate Efficacy at 24 Weeks and to Assess the Long Term Safety, Tolerability and Efficacy up to 3 Years in Subjects With Active Psoriatic Arthritis
Brief Title: 24 Week Efficacy and 3-year Safety and Efficacy of Secukinumab in Active Psoriatic Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F2318; 2013-004002-25 (EudraCT Number)
Record Dates: First submitted 2013-11-07; First posted 2013-11-21 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic arthritis; AIN457; PsA; ACR; CASPAR; PASDAS; secukinumab; autoinjector
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Secukinumab (AIN457) 150 mg s.c. (Experimental): 1 s.c. Secukinumab 150 mg autoinjector at Baseline, Weeks 1, 2, 3, 4, followed by dosing every four weeks starting at Week 4.
  Interventions: Biological: Secukinumab
- Secukinumab (AIN457) 300 mg s.c. (Experimental): 2 s.c. Secukinumab 150 mg autoinjector at Baseline, Weeks 1, 2, 3, 4, followed by dosing every four weeks starting at Week 4.
  Interventions: Biological: Secukinumab
- Placebo (Placebo Comparator): Matching Placebo at Baseline, Weeks 1, 2, 3, 4, followed by dosing every four weeks starting at Week 4.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Secukinumab — Secukinumab 150 mg provided in a 1 mL autoinjector (1 autoinjector for 150 mg dose, 2 autoinjectors for 300 mg dose)
  Other Names: Secukinumab 150 mg; Secukinumab 300 mg
  Arms: Secukinumab (AIN457) 150 mg s.c.; Secukinumab (AIN457) 300 mg s.c.
Biological: Placebo — Secukinumab placebo provided in 1 mL autoinjector
  Arms: Placebo

SUMMARY:
The purpose of this study is to provide 24 - 52 week efficacy, safety and tolerability data, and up to 3-year efficacy, safety and tolerability data in subjects with active Psoriatic Arthritis despite current or previous nonsteroidal anti-inflammatory drug (NSAID), disease-modifying antirheumatic drug (DMARD) therapy and/or previous anti-tumor necrosis factor alpha (TNFα) therapy.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Psoriatic Arthritis (PsA) classified by ClASsification criteria for Psoriatic ARthritis (CASPAR) criteria.
* Rheumatoid factor and anti-cyclic citrullinated peptide (CCP) antibodies negative.
* Diagnosis of active plaque psoriasis or nail changes consistent with psoriasis.
* Inadequate control of symptoms with NSAID.

Exclusion Criteria:

* Chest X-ray or chest magnetic resonance imaging (MRI) with evidence of ongoing infectious or malignant process.
* Subjects taking high potency opioid analgesics.
* Previous exposure to secukinumab or other biologic drug directly targeting interleukin-17 (IL-17) or IL-17 receptor.
* Ongoing use of prohibited psoriasis treatments / medications.
* Subjects who have ever received biologic immunomodulating agents except for those targeting TNFα.
* Previous treatment with any cell-depleting therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2015-05-27 (Actual); Study Completion 2018-03-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (72):
- United States (12):
  - Novartis Investigative Site, Aventura, Florida
  - Novartis Investigative Site, Palm Harbor, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Bowling Green, Kentucky
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Freehold, New Jersey
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, Mesquite, Texas
  - Novartis Investigative Site, Wenatchee, Washington
- Australia (4):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Maroochydore, Queensland
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Malvern East, Victoria
- Bulgaria (2):
  - Novartis Investigative Site, Sofia
  - Novartis Investigative Site, Veliko Tarnovo
- Canada (4):
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Czechia (3):
  - Novartis Investigative Site, Bruntál, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Uherské Hradiště, Czech Republic
- Germany (10):
  - Novartis Investigative Site, Aachen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Chemnitz
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Gommern
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Zerbst
- Italy (7):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Catania, CT
  - Novartis Investigative Site, Genova, GE
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Reggio Emilia, RE
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Verona, VR
- Netherlands (3):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Heerlen
  - Novartis Investigative Site, Rotterdam
- Puerto Rico (2):
  - Novartis Investigative Site, Caguas
  - Novartis Investigative Site, Ponce
- Russia (7):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saratov
  - Novartis Investigative Site, Sestroretsk
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Spain (4):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Santander, Cantabria
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
- Switzerland (2):
  - Novartis Investigative Site, Fribourg
  - Novartis Investigative Site, Sankt Gallen
- United Kingdom (12):
  - Novartis Investigative Site, London, England
  - Novartis Investigative Site, Salford, Manchester
  - Novartis Investigative Site, Cannock, Staffordshire
  - Novartis Investigative Site, Stoke-on-Trent, Staffordshire
  - Novartis Investigative Site, Barnsley
  - Novartis Investigative Site, Eastbourne
  - Novartis Investigative Site, Harrogate
  - Novartis Investigative Site, Hull
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Torquay
  - Novartis Investigative Site, Tyne and Wear

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Mease PJ, Warren RB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, McInnes IB. Comparative Effectiveness of Bimekizumab and Secukinumab in Patients with Psoriatic Arthritis at 52 Weeks Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Jun;11(3):817-828. doi: 10.1007/s40744-024-00652-7. Epub 2024 Mar 6. PMID 38446397
- [Derived] Pournara E, Kormaksson M, Nash P, Ritchlin CT, Kirkham BW, Ligozio G, Pricop L, Ogdie A, Coates LC, Schett G, McInnes IB. Clinically relevant patient clusters identified by machine learning from the clinical development programme of secukinumab in psoriatic arthritis. RMD Open. 2021 Nov;7(3):e001845. doi: 10.1136/rmdopen-2021-001845. PMID 34795065
- [Derived] Coates LC, Wallman JK, McGonagle D, Schett GA, McInnes IB, Mease PJ, Rasouliyan L, Quebe-Fehling E, Asquith DL, Fasth AER, Pricop L, Gaillez C. Secukinumab efficacy on resolution of enthesitis in psoriatic arthritis: pooled analysis of two phase 3 studies. Arthritis Res Ther. 2019 Dec 4;21(1):266. doi: 10.1186/s13075-019-2055-z. PMID 31801620
- [Derived] Deodhar A, Gladman DD, McInnes IB, Spindeldreher S, Martin R, Pricop L, Porter B, Safi J Jr, Shete A, Bruin G. Secukinumab Immunogenicity over 52 Weeks in Patients with Psoriatic Arthritis and Ankylosing Spondylitis. J Rheumatol. 2020 Apr;47(4):539-547. doi: 10.3899/jrheum.190116. Epub 2019 Jun 15. PMID 31203228
- [Derived] Nash P, Mease PJ, McInnes IB, Rahman P, Ritchlin CT, Blanco R, Dokoupilova E, Andersson M, Kajekar R, Mpofu S, Pricop L; FUTURE 3 study group. Efficacy and safety of secukinumab administration by autoinjector in patients with psoriatic arthritis: results from a randomized, placebo-controlled trial (FUTURE 3). Arthritis Res Ther. 2018 Mar 15;20(1):47. doi: 10.1186/s13075-018-1551-x. PMID 29544534

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were randomized to 1 of 3 treatment arms (1:1:1) and planned to be treated for 156 weeks. Placebo non-responders had the option to be re-randomized at Week 16 and placebo responders had the option to be re-randomized at Week 24. Thus, of the 137 original placebo patients 64 were re-randomized to AIN457 150 mg and 65 to AIN457 300 mg.
Pre-assignment Details: A screening period (SCR) running up to 10 weeks before randomization was used to assess eligibility.
Groups:
- AIN457 150 mg: 1 s.c. Secukinumab 150 mg autoinjector at Baseline, Weeks 1, 2, 3, 4, followed by dosing every four weeks starting at Week 4.
- AIN457 300 mg: 2 s.c. Secukinumab 150 mg autoinjector at Baseline, Weeks 1, 2, 3, 4, followed by dosing every four weeks starting at Week 4.
- Placebo_AIN457 150 mg: Placebo switch to Secukinumab/AIN457 150 mg
- Placebo_AIN457 300 mg: Placebo switch to Secukinumab/AIN457 300 mg
- Placebo Not Rerandomized: Matching Placebo at Beseline, Weeks 1, 2, 3, 4, followed by dosing every four weeks starting at Week 4.
Period: Overall Study
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo_AIN457 150 mg | Placebo_AIN457 300 mg | Placebo Not Rerandomized
Started (All randomized patients were included in the Full Analysis Set (FAS) and Safety Set (SAF).) | 138 | 139 | 64 | 65 | 8
Completed (Completed Week 156) | 91 | 102 | 45 | 49 | 0
Not Completed | 47 | 37 | 19 | 16 | 8
Not completed — Adverse Event | 10 | 15 | 4 | 5 | 4
Not completed — Lack of Efficacy | 11 | 11 | 7 | 4 | 2
Not completed — Lost to Follow-up | 5 | 2 | 0 | 1 | 1
Not completed — Physician Decision | 4 | 1 | 0 | 1 | 0
Not completed — Pregnancy | 0 | 1 | 0 | 0 | 0
Not completed — Technical Problems | 3 | 1 | 3 | 1 | 0
Not completed — Subject Guardian Decision | 11 | 6 | 4 | 4 | 1
Not completed — Death | 3 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Matching Placebo at Beseline, Weeks 1, 2, 3, 4, followed by dosing every four weeks starting at Week 4.
- Total: Total of all reporting groups
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo | Total
Number analyzed (Participants) | 138 | 139 | 137 | 414
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 126 | 123 | 118 | 367
  >=65 years | 12 | 16 | 19 | 47
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 72 | 78 | 227
  Male | 61 | 67 | 59 | 187
Race/Ethnicity, Customized [Number; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 2 | 3 | 4 | 9
  White | 129 | 130 | 133 | 392
  Other | 5 | 6 | 0 | 11

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Achieving American College of Rheumatology 20 (ACR20) Response Criteria on Secukinumab Versus Placebo at Week 24
Description: A patient will be considered as improved according the ACR20 criteria if she/he has at least 20% decrease in the swollen and tender joint count, and at least 20% improvements in 3 of the following 5 criteria: physical disability on the Health Assessment Questionnaire; pain score on a visual analog scale; patient global assessment; physician global assessment; and acute phase reactant [either erythrocyte sedimentation rate (ESR) or high sensitivity C-reactive protein (hsCRP)]
Time Frame: Week 24
Population: The Full Analysis Set (FAS) based on Primary Analysis, which consisted of all participants with an observed value, was considered.
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 138 | 139 | 137
Participants | 58 | 67 | 22

2. Secondary Outcome: Proportion of Patients Achieving American College of Rheumatology 50 (ACR50) Response Criteria on Secukinumab Versus Placebo at Week 24
Description: A patient will be considered as improved according the ACR50 criteria if she/he has at least 50% decreases in the swollen and tender joint count, and at least 50% improvements in 3 of the following 5 criteria: physical disability on the Health Assessment Questionnaire; pain score on a visual analog scale; patient global assessment; physician global assessment; and acute phase reactant [either erythrocyte sedimentation rate (ESR) or high sensitivity C-reactive protein (hsCRP)]
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 138 | 139 | 137
Participants | 26 | 48 | 12

3. Secondary Outcome: Change From Baseline in Disease Activity Score for 28 Joints (DAS28-CRP) (Utilizing hsCRP) in Subjects Treated With Secukinumab Versus Placebo at Week 24
Description: DAS28-CRP is a measure of disease activity based on 28-Swollen and Tender Joint Count [proximal interphalangeal joints (10 joints) metacarpophalangeal joints (10) wrists (2) elbows (2) shoulders (2) knees (2)], CRP, and the Patient's Global Assessment of disease activity. Values range from 2.0 to 10.0 where higher values mean a higher disease activity. DAS28-CRP < 2.6 is interpreted as remission.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 138 | 139 | 137
Unit on a scale | -1.24 (0.095) | -1.56 (0.093) | -0.64 (0.127)

4. Secondary Outcome: Proportion of Subjects Achieving a Psoriatic Area and Severity Index 75 (PASI75) Response in Subjects on Secukinumab Versus Placebo at Week 24
Description: PASI takes into account the extent of the disease, as well as the severity of erythema, scaling, and thickness in different body areas affected by psoriasis. A PASI75 represents an improvement in the PASI score of at least 75% as compared with baseline.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 68 | 62 | 59
Participants | 34 | 29 | 6

5. Secondary Outcome: Change From Baseline in Physical Function Component of the Short-form Health Survey (SF-36-PCS) in Subjects Treated With Secukinumab Versus Placebo at Week 24
Description: SF-36 is a 36 item questionnaire which measures Quality of Life across eight domains, which are both physically and emotionally based. Two overall summary scores, the Physical Component Summary (PCS) and Mental Component Summary (MCS) can be computed. In this study, SF-36 PCS is used to assess improvement from baseline of at least one dose of secukinumab versus placebo. The SF-36 is a validated instrument measuring health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores (1) physical component summary=physical functioning, role-physical, bodily pain, and general health. There is no total overall score; scoring is done for both subscores and summary scores. For subscores and summary scores, 0 =worst score (or quality of life) and 100=best score. Change from Baseline= post-Baseline - Baseline value.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 138 | 139 | 137
Unit on a scale
  Mental Component Summary (MCS): number analyzed (Participants) | 125 | 130 | 42
  Mental Component Summary (MCS) | 1.68 (0.837) | 4.41 (0.822) | -0.10 (1.142)
  Physical Component Summary (PCS): number analyzed (Participants) | 125 | 130 | 42
  Physical Component Summary (PCS) | 3.42 (0.600) | 6.46 (0.590) | 2.94 (0.830)

6. Secondary Outcome: Percentage of Subjects Achieving a Psoriatic Area and Severity Index 90 (PASI90) Response in Subjects Treated With Secukinumab Versus Placebo at Week 24
Description: PASI takes into account the extent of the disease, as well as the severity of erythema, scaling, and thickness in different body areas affected by psoriasis. A PASI90 represents an improvement in the PASI score of at least 90% as compared with baseline.
Time Frame: Week 24
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 68 | 62 | 59
Participants | 25 | 21 | 4

7. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI Score) in Subjects Treated With Secukinumab Versus Placebo at Week 24
Description: The HAQ measures physical disability and functional status. It has 4 dimensions: disability, pain, drug side effects and dollar costs. In this trial, only the disability dimension was used. The disability dimension consists of 20 multiple choice items concerning difficulty in performing 8 common activities of daily living; dressing and grooming, arising, eating, walking, reaching, personal hygiene, gripping and activities. Participants choose from four response categories: 0 (without any difficulty), 1 (with some difficulty), 2 (with much difficulty) and 3 (unable to do). Within each of the 8 categories, only the item indicating the most severe impairment contributes to the category score. The HAQ score is calculated by summing the computed scores for each category and dividing by the number of categories answered. It ranges from 0 (without any difficulty) to 3 (unable to do). A negative change from baseline indicates improvement.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 138 | 139 | 137
Unit on a scale | -0.27 (0.043) | -0.38 (0.042) | -0.17 (0.055)

8. Secondary Outcome: Proportion of Patients With Dactylitis at Week 24 in the Subset of Patients Who Had Dactylitis at Baseline
Description: The presence of dactylitis was assessed by dactylitis count (number of fingers and toes with dactylitis, with a range of 0-20). If dactylitis is present with any finger or toe, the patient is counted as a patient with dactylitis.
Time Frame: Week 24
Population: The Dactylitis subset of the Full Analysis Set (FAS) based on Primary Analysis, which consisted of all participants with an observed value at Baseline and post-basline, was considered.
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 36 | 46 | 36
Participants | 22 | 24 | 31

9. Secondary Outcome: Proportion of Patients With Enthesitis at Week 24 in the Subset of Patients Who Had Enthesitis at Baseline
Description: The presence of Enthesitis was assessed using a validated enthesitis index that uses 6 sites for evaluation of enthesitis: lateral epicondyle humerus L + R, proximal achilles L + R and medial condyle femur. If enthesitis is present at any of the 6 sites, the subject is counted as a subject with enthesitis.
Time Frame: Week 24
Population: The Enthesitis subset of the Full Analysis Set (FAS) based on Primary Analysis, which consisted of all participants with an observed value at Baseline and post-basline, was considered.
Measure: Count of Participants; unit: Participants
Arm/Group | AIN457 150 mg | AIN457 300 mg | Placebo
Number analyzed (Participants) | 95 | 88 | 98
Participants | 60 | 53 | 83

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Event (AE), Serious Adverse Event (SAE) and Deaths by Primary System Organ Class (SOC)
Description: Analysis of frequencies for treatment emergent Adverse Event (AE), Serious Adverse Event (SAE) and Deaths by primary System Organ Class (SOC).
Time Frame: From first dose of study treatment to last study visit, up to 3 years
Population: Safety Set, based on Final Analysis. All subjects who took at least one dose of study treatment during the treatment period. A subject with multiple adverse events within a primary system organ class was counted only once in the total row. Deaths up to 28 days after the last dose are included. Only descriptive analysis done.
Measure: Count of Participants; unit: Participants
Groups:
- Any AIN457 150 mg: Any patients exposed to AIN457 150 mg
- Any AIN457 300 mg: Any patients exposed to AIN457 300 mg
- Any AIN457: Any patients exposed to AIN457
Arm/Group | Any AIN457 150 mg | Any AIN457 300 mg | Any AIN457 | Placebo
Number analyzed (Participants) | 202 | 284 | 406 | 137
Participants
  AEs by Primary System Organ Class (SOC) | 176 | 230 | 363 | 81
  SAEs by Primary System Organ Class (SOC) | 42 | 35 | 76 | 9
  Deaths by Primary System Organ Class (SOC) | 4 | 0 | 4 | 0

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) are reported in this record from date of First Patient First Treatment (FPFT) until end of treatment exposure, up to 156 weeks, + 84 days safety follow-up.
Groups:
- Any AIN457 150 mg: 1 s.c. Secukinumab 150 mg autoinjector at Baseline, Weeks 1, 2, 3, 4, followed by dosing every four weeks starting at Week 4.
- Any AIN457 300 mg: 2 s.c. Secukinumab 150 mg autoinjector at Baseline, Weeks 1, 2, 3, 4, followed by dosing every four weeks starting at Week 4.
Arm/Group | Any AIN457 150 mg | Any AIN457 300 mg | Any AIN457 | Placebo
All-Cause Mortality (participants affected / at risk) | 4/202 | 0/284 | 4/406 | 0/137
Serious Adverse Events (participants affected / at risk) | 42/202 | 35/284 | 76/406 | 9/137
Other Adverse Events (participants affected / at risk) | 153/202 | 201/284 | 320/406 | 65/137
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg (N=202) | Any AIN457 300 mg (N=284) | Any AIN457 (N=406) | Placebo (N=137)
Lymphadenitis (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1 | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 1 | 0
Angina unstable (Cardiac disorders) | 0 | 1 | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 0 | 1 | 1 | 0
Arrhythmia (Cardiac disorders) | 0 | 1 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 1 | 2 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 1 | 0 | 1 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 1 | 0
Cardiogenic shock (Cardiac disorders) | 1 | 0 | 1 | 0
Diastolic dysfunction (Cardiac disorders) | 0 | 1 | 1 | 0
Left ventricular hypertrophy (Cardiac disorders) | 0 | 1 | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 0 | 1 | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 2 | 0
Sudden hearing loss (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Vestibular disorder (Ear and labyrinth disorders) | 1 | 0 | 1 | 0
Cataract (Eye disorders) | 1 | 1 | 2 | 0
Retinal detachment (Eye disorders) | 1 | 0 | 1 | 0
Anal prolapse (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Inflammatory bowel disease (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Asthenia (General disorders) | 1 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 1 | 0
Biliary dyskinesia (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Abscess jaw (Infections and infestations) | 0 | 1 | 1 | 0
Abscess of salivary gland (Infections and infestations) | 0 | 1 | 1 | 0
Arthritis bacterial (Infections and infestations) | 0 | 1 | 1 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 2 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 2 | 2 | 0
Eczema infected (Infections and infestations) | 0 | 1 | 1 | 0
Enterococcal sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 1 | 0
Infectious mononucleosis (Infections and infestations) | 0 | 0 | 0 | 1
Joint abscess (Infections and infestations) | 1 | 0 | 1 | 0
Periodontitis (Infections and infestations) | 0 | 1 | 1 | 0
Pneumonia (Infections and infestations) | 3 | 1 | 4 | 0
Staphylococcal infection (Infections and infestations) | 1 | 0 | 1 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 2 | 0
Wound infection (Infections and infestations) | 0 | 1 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Cardiac valve rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Ligament rupture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 2 | 2 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Sternal fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Traumatic arthrosis (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Weight decreased (Investigations) | 0 | 1 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 4 | 6 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Follicular thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Invasive papillary breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Lip squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Ovarian cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Phyllodes tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 1 | 0
Cerebral ischaemia (Nervous system disorders) | 1 | 0 | 1 | 0
Coma (Nervous system disorders) | 1 | 0 | 1 | 0
Depressed level of consciousness (Nervous system disorders) | 1 | 0 | 1 | 0
Facial paresis (Nervous system disorders) | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 1 | 0 | 1 | 0
Hemiplegia (Nervous system disorders) | 1 | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 1 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0 | 1 | 0
Quadriparesis (Nervous system disorders) | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 1 | 1 | 0
Device dislocation (Product Issues) | 1 | 0 | 1 | 1
Device loosening (Product Issues) | 1 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 1 | 0
Sopor (Psychiatric disorders) | 1 | 0 | 1 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 1 | 2 | 0
Urethral stenosis (Renal and urinary disorders) | 1 | 0 | 1 | 0
Cystocele (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Ovarian cyst torsion (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Rectocele (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Uterovaginal prolapse (Reproductive system and breast disorders) | 1 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0
Circulatory collapse (Vascular disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 1 | 1
Peripheral artery thrombosis (Vascular disorders) | 1 | 0 | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg (N=202) | Any AIN457 300 mg (N=284) | Any AIN457 (N=406) | Placebo (N=137)
Anaemia (Blood and lymphatic system disorders) | 6 | 3 | 9 | 0
Palpitations (Cardiac disorders) | 5 | 4 | 9 | 0
Abdominal pain (Gastrointestinal disorders) | 4 | 8 | 12 | 0
Abdominal pain upper (Gastrointestinal disorders) | 10 | 9 | 17 | 2
Constipation (Gastrointestinal disorders) | 5 | 6 | 11 | 1
Diarrhoea (Gastrointestinal disorders) | 20 | 19 | 39 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 6 | 12 | 1
Mouth ulceration (Gastrointestinal disorders) | 6 | 2 | 8 | 0
Nausea (Gastrointestinal disorders) | 12 | 18 | 30 | 7
Vomiting (Gastrointestinal disorders) | 4 | 3 | 7 | 4
Fatigue (General disorders) | 16 | 10 | 26 | 2
Injection site erythema (General disorders) | 1 | 2 | 3 | 3
Non-cardiac chest pain (General disorders) | 5 | 2 | 7 | 1
Oedema peripheral (General disorders) | 1 | 6 | 7 | 0
Bronchitis (Infections and infestations) | 11 | 23 | 34 | 6
Conjunctivitis (Infections and infestations) | 4 | 9 | 13 | 1
Cystitis (Infections and infestations) | 6 | 5 | 11 | 1
Ear infection (Infections and infestations) | 1 | 6 | 7 | 1
Gastroenteritis (Infections and infestations) | 10 | 10 | 20 | 1
Influenza (Infections and infestations) | 12 | 16 | 26 | 3
Lower respiratory tract infection (Infections and infestations) | 6 | 4 | 10 | 0
Nasopharyngitis (Infections and infestations) | 44 | 63 | 105 | 16
Oral candidiasis (Infections and infestations) | 5 | 6 | 11 | 0
Oral herpes (Infections and infestations) | 4 | 8 | 12 | 1
Otitis media (Infections and infestations) | 0 | 6 | 6 | 0
Pharyngitis (Infections and infestations) | 4 | 8 | 12 | 1
Respiratory tract infection (Infections and infestations) | 6 | 13 | 18 | 0
Respiratory tract infection viral (Infections and infestations) | 0 | 5 | 5 | 3
Rhinitis (Infections and infestations) | 5 | 7 | 12 | 0
Sinusitis (Infections and infestations) | 10 | 12 | 22 | 4
Tonsillitis (Infections and infestations) | 4 | 14 | 18 | 1
Upper respiratory tract infection (Infections and infestations) | 27 | 35 | 61 | 7
Urinary tract infection (Infections and infestations) | 13 | 20 | 31 | 2
Viral upper respiratory tract infection (Infections and infestations) | 5 | 4 | 9 | 1
Fall (Injury, poisoning and procedural complications) | 5 | 11 | 15 | 1
Limb injury (Injury, poisoning and procedural complications) | 8 | 2 | 10 | 1
Alanine aminotransferase increased (Investigations) | 11 | 6 | 17 | 1
Aspartate aminotransferase increased (Investigations) | 8 | 3 | 11 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 6 | 3 | 9 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 1 | 6 | 7 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 23 | 40 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 7 | 8 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 24 | 41 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5 | 4 | 9 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 6 | 6 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 2 | 4 | 3
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 14 | 14 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 5 | 10 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 20 | 21 | 41 | 5
Dizziness (Nervous system disorders) | 7 | 3 | 10 | 2
Headache (Nervous system disorders) | 18 | 18 | 36 | 7
Sciatica (Nervous system disorders) | 4 | 5 | 9 | 0
Depression (Psychiatric disorders) | 5 | 3 | 8 | 0
Haematuria (Renal and urinary disorders) | 0 | 4 | 4 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 17 | 12 | 29 | 6
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 | 15 | 25 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 11 | 15 | 26 | 3
Rash (Skin and subcutaneous tissue disorders) | 5 | 2 | 7 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 6 | 7 | 1
Hypertension (Vascular disorders) | 11 | 15 | 26 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.